CLINICAL TRIAL: NCT00441194
Title: To Compare the Octopus 311 and the Humphrey Field Analyzer 700 Series With Respect to Reliability, Reproducibility, Test Duration, Patient Preference, Technician Preference.
Brief Title: To Compare the Octopus 311 and the Humphrey Field Analyzer 700 Series
Status: Terminated | Type: Observational
Why Stopped: Study terminated due to resources
Sponsor: Haag Streit USA (Industry)
Other Study IDs: HSOCT001
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Visual Field
Keywords: Perimetry; Visual Field; Octopus
MeSH Terms: interventions — Visual Field Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Visual Field (Octopus 311 and the HFA 700 series)

SUMMARY:
To compare the Octopus 311 and the HFA 700 series

DETAILED DESCRIPTION:
To compare the Octopus 311 and the HFA 700 series to evaluate reliability, reproducibility, test duration, patient preference and technician preference.

ELIGIBILITY:
Inclusion Criteria:

* Prior Visual Field

Exclusion Criteria:

* Scotopic pupil less than 3 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2006-11; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Powers, O.D., Principal Investigator — American, Virginia and Northern Virginia Optometric Associations
Locations (1):
- Capital Eye Consultants, Fairfax, Virginia, United States